CLINICAL TRIAL: NCT01209559
Title: A Comparative Study of the Air-Q ILA and the ILMA for Ventilation and Intubation
Status: Withdrawn | Type: Observational
Why Stopped: Study never initiated.
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Orlando Hung, MD FRCPC, Nova Scotia Health Authority
Other Study IDs: CDHA-RS/2011-156
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Airway Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- air-Q Intubating Laryngeal Airway
- LMA FastrachTM or ILMA

SUMMARY:
The objective of this study is to determine if the glottic view obtained with the air-Q Intubating Laryngeal Airway (air-Q ILA, Cookgas LLC®, Mercury Medical®, Clearwater, FL, USA) is better than that obtained with the traditionally used intubating laryngeal mask airway (LMA FastrachTM or ILMA, LMA North America Inc., San Diego, CA). The study will also compare effectiveness of ventilation.

ELIGIBILITY:
Inclusion Criteria:

* healthy ASA class I and II patients scheduled for elective surgery under general anesthesia requiring the use of the LMA

Exclusion Criteria:

* history of acid reflux,
* a BMI ≥ 40kg.m-2,
* require endotracheal intubation,
* have predictors of difficult intubation,
* not candidates for insertion of an ILMA or LMA, including a mouth opening of less than 2.5 cm,
* cannot consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy ASA class I and II patients scheduled for elective surgery under general anesthesia requiring the use of the LMA.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada